CLINICAL TRIAL: NCT00307528
Title: A Study to Evaluate the Safety, Reactogenicity & Immunogenicity of the GSK Biologicals Candidate Pneumococcal Vaccine Without or With Adjuvant, Administered at 2 Different Concentrations, in Healthy Elderly Subjects
Brief Title: Safety and Efficacy Study of Investigational Pneumococcal Vaccine in Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100409; 100463 (Other: GSK); 100464 (Other: GSK)
Record Dates: First submitted 2006-03-06; First posted 2006-03-28 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Prophylaxis Invasive Pneumococcal Diseases and Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- Group A (Active Comparator)
  Interventions: Biological: Pneumovax 23™
- Group B (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK513026
- Group C (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK513026
- Group D (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK513026
- Group E (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK513026
- Group F (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK513026

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK513026 — Two-dose intramuscular injection. Five different formulations, each administered to one Group
  Arms: Group B; Group C; Group D; Group E; Group F
Biological: Pneumovax 23™ — Single dose intramuscular injection.
  Arms: Group A

SUMMARY:
As the licensed Pneumovax 23™ vaccine is not always satisfactory in elderly subjects, the safety and the immune response of the new investigational pneumococcal protein vaccine is evaluated in healthy elderly population.

DETAILED DESCRIPTION:
Since influenza vaccination is recommended in the age range of the study population, Fluarix™ (GlaxoSmithKline Biologicals) vaccine will be offered free of charge during the study period (for 3 consecutive years starting from September 2004), to be used by Investigators according to national vaccination schedule/practice.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria

* Subjects who the investigator believes will comply with the requirements of the protocol
* A male or female ≥ 65 years at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion criteria

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Use of any anticoagulants.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 2 weeks of the first dose of vaccines.
* Previous vaccination against Streptococcus pneumoniae.
* Bacterial pneumonia within 3 years prior to 1st vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Current serious neurologic or mental disorders.
* Currently smoking > 25 cigarettes per day.
* Inflammatory processes such as known chronic active infections
* All malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* History of administration of an experimental vaccine containing MPL or QS21.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, at the discretion of the investigator.
* History of chronic alcohol consumption and/or intravenous drug abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 146 (Actual)
Dates: Start 2004-01-20 (Actual); Primary Completion 2005-03-30 (Actual); Study Completion 2005-03-30 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship of any solicited local and general signs and symptoms. | During a 7-day follow up period after each vaccine dose.
Occurrence, intensity and relationship to vaccination of unsolicited local and general signs and symptoms. | During a 30-day follow up period after each vaccine dose.
Occurrence of all serious adverse events (SAE). | During the entire study period.
Anti- PhtD antibody concentration | One month after the first injection
Anti-PhtD antibody concentration. | One month after 2 injections

SECONDARY OUTCOMES:
Number and percentage of subjects with normal or abnormal values for biochemical assessments and for haematological analysis. | At each scheduled time point (month 0, 1, 3, 12, 24 and 36).
Anti- PhtD antibody concentration. | At 12, 24 and 36 months after the first vaccination.
Anti-PhtD antibody avidity. | At month 0, 1 and 3.
Evaluation of protection afforded by passive transfer of anti PhtD antibodies sera pooled from all individuals. | At month 0, 1 and 3.
Frequency of PhtD specific plasma cells generated by in vitro cultivated memory B-cells, in a subset of subjects. | At month 0, 1, 3, 12.
Frequency of CD4 and/or CD8 T cells that produce cytokines (IL-2, IL-4, IFNg, CD40L and/or GM-CSF, and TNFα), upon PhtD re-stimulation in vitro, to evaluate the T-cell response, in a subset of subjects. | At month 0, 1, 3, 12.
Anti-polysaccharide total IgG concentration in Group A for all vaccine pneumococcal serotypes | At month 0, 1, 12, 24 and 36.
Anti-PS antibody avidity for 5 serotypes in Group A. | At month 0 and 1.
Deposition of complement components on the surface of different bacterial strains 3 strains (GSK/CDC, OPA, isogenic TIGR4) of 5 serotypes in Group A. | At month 0 and 1.
Opsonophagocytic activity titres in Group A to all vaccine pneumococcal serotypes | At month 0, 1 and 12.
Frequency of PS-specific plasma cells generated by in vitro cultivated memory B-cells in Group A in a subset of subjects. | At month 0 and month 1.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=1980

REFERENCES:
- [Derived] Leroux-Roels I, Devaster JM, Leroux-Roels G, Verlant V, Henckaerts I, Moris P, Hermand P, Van Belle P, Poolman JT, Vandepapeliere P, Horsmans Y. Adjuvant system AS02V enhances humoral and cellular immune responses to pneumococcal protein PhtD vaccine in healthy young and older adults: randomised, controlled trials. Vaccine. 2015 Jan 15;33(4):577-84. doi: 10.1016/j.vaccine.2013.10.052. Epub 2013 Oct 29. PMID 24176494